CLINICAL TRIAL: NCT02748460
Title: Prospective, Multi-national, Multicentre, Non-interventional Study to Evaluate the Long Term Safety of Esmya, in Particular Endometrial Safety, and the Current Prescription and Management Patterns of Esmya in a Long Term Treatment Setting.
Brief Title: Non-interventional Study to Evaluate Long Term Safety, Prescription Management Patterns of Esmya in a Long Term Setting
Acronym: Premium
Status: Completed | Type: Observational
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Other Study IDs: PGL14-001 (PREMIUM)
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Esmya: Any patient who was confirmed as receiving one dose of Esmya

SUMMARY:
This is a multi-centre, multinational, prospective, non-interventional study in females with a diagnosis of moderate to severe uterine fibroids, and for whom a treatment with Esmya in a long term manner is planned, and in subjects who were previously exposed to UPA in the long term Phase III studies.

DETAILED DESCRIPTION:
This is a multi-centre, multinational, prospective, non-interventional study in females with a diagnosis of moderate to severe uterine fibroids, and for whom a treatment with Esmya in a long term manner is planned, and in subjects who were previously exposed to UPA in the long term Phase III studies. It is planned to enrol approximately 1,500 patients. Consecutive, eligible, patients will be invited to enrol from approximately 100-150 European Union (EU) clinical practice sites in approximately 15 countries. Patients will be followed for an observation period of 60 months (5 years) from treatment start. Investigators are to manage and treat patients according to their standard medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult women of reproductive age with a diagnosis of moderate to severe symptoms of uterine fibroids who are not eligible for surgery and for whom a intermittent treatment with Esmya in a long term manner (at least 2 courses), is planned or subjects who were exposed to UPA 5 or 10 mg during long term Phase III trials PGL09-027 (PEARL III extension, including patients (PEARL extension 2)) or PGL11-006 (PEARL IV), and
* Patient is willing and able to attend visits which are scheduled by her treating physician for the regular follow-up, provide the required medical data, and
* Patient has personally signed and dated the informed consent document indicating that she has been informed of all pertinent aspects of the study.

Exclusion criteria:

* Patient is prescribed Esmya for pre-operative treatment
* Patient has a contraindication to receive Esmya as per SmPC
* Patient is using an investigational drug/therapy or has discontinued the use of an investigational drug/therapy within 30 days prior to study enrolment,
* Patient has hypersensitivity to the active substance of Esmya or to one of its excipients,
* Not applicable to long term phase III previous subjects who are not planning to receive Esmya during this study:

  * Patient is pregnant or plans to become pregnant within the next 12 months from treatment start,
  * Patient is breastfeeding,
  * Patient has genital bleeding of unknown aetiology or not due to uterine fibroids,
  * Patient has been diagnosed with uterine, cervical, ovarian or breast cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will include women with moderate to severe symptoms of uterine fibroids, and for whom a treatment with Esmya in a long term manner is planned, and subjects who were previously exposed to UPA 5 or 10 mg in Long Term Phase III clinical trials PGL09-027 (PEARL III extension; including patients of PGL11-024 (PEARL extension 2)), or PGL11-006 (PEARL IV).
Sampling Method: Non-Probability Sample
Enrollment: 1527 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Assessment of long term safety: Occurrence of gynaecological AEs, SAEs, non-serious ADRs, AEs leading to ESMYA treatment discontinuation | Patients will be followed from baseline up to 60 months
  Occurrence of gynaecological AEs, SAEs, non-serious ADRs, AEs leading to ESMYA treatment discontinuation

SECONDARY OUTCOMES:
Assessment of Prescription pattern of Esmya in standard medical practice | Patients will be followed from baseline up to 60 months
  Esmya use in patients

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Arriagada, Study Director — PregLem SA
Locations (115):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Regional De La Citadelle, Liège
  - Clinique Universitaire de Mont Godinne, Yvoir
- Czechia (7):
  - Dr Dvorak, Brno
  - Gyn-Porodnicka Klinika Fn Brno, Brno
  - Gyn -Fsro, Králová
  - G-Centrum Olomouc S.R.O., Olomouc
  - Private Practice 2, Prague
  - Private Practice, Prague
  - Uherskohradistska Nemocnice A.S, Uherské Hradiště
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Gastroenheden Herlev-Gentofte, Herlev
- France (5):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier de Bethune, Béthune
  - Groupement Hospitalier Universitaire Sud CHU Bicetre, Le Kremlin-Bicêtre
  - Hopital Bichat - Claude-Bernard, Paris
  - Centre Hospitalier Regional Universitaire de Tours (CHRU de Tours) - Hopital Bretonneau, Tours
- Germany (26):
  - Private practice, Aachen
  - Klinikum Bayreuth GmbH, Bayreuth
  - Charite -Universitatsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Praxis fuer Gynaekologie & Geburtshilfe Prof. Dr. Dr. A. Ebert, Berlin
  - Gynakologische Praxis Klinik, Bonn
  - PAN-Klinik am Neumarkt-Gemeinschaftspraxis fur Urologie, Cologne
  - Gemeinschaftspraxis der Frauenarztpraxis, Deggendorf
  - Private Practice, Dortmund
  - Private Practice, Frankfurt
  - Frauenarztpraxis, Frankfurt am Main
  - Hellweg gynakologie/DOCX, Geseke
  - Universitaetsklinikum Giessen und Marburg GmbH, Giessen
  - Frauenarztpraxis Gluckstadt, Glückstadt
  - Frauenarzt Bergedorf, Hamburg
  - Frauenarztpraxis Wandsbek, Hamburg
  - Praxisklinik Harburg, Hamburg
  - Private Practice, Hamburg
  - Unversitaetsklinikum Hamburg Eppendorf - Klinik und Poliklinik fur Gynakologie, Hamburg
  - Private practice, Ilsede
  - Frauenarztpraxis, Köthen
  - Medplus Krefeld, Krefeld
  - Endoskopie Und Endometriose-Zentrum Munchen, München
  - Private Practice, Plöcking
  - Private practice, Ribnitz-Damgarten
  - Private Practice, Stolberg
  - Ammerland Klinik GmbH, Westerstede
- Hungary (6):
  - Rethy Pal Hospital-Clinic Bekescsaba, Békéscsaba
  - Robert Karoly Maganklinika, Budapest
  - Szent Anna Privat Surgery-Szent Anna Magae¡nrendela, Debrecen
  - Josa Andras County Teaching Hospital, Nyíregyháza
  - Szegedi Tudomanyegyetem, Szuleszeti es Nogyogyaszati Klinika, Szeged
  - Csongrad Megyei Dr. Bugyi Istvan Korhaz, Szentes
- Italy (9):
  - Woman's Health Sciences Department, Gynecologic Section, Hsopital G. Salesi- Polytechnic University of Marche, Ancona
  - University of Bari Policlinico, Bari
  - Azienda Usl Di Bologna, Bologna
  - Policlinico S. Orsola Malpighi, Bologna
  - A.O.Spedali Civili di Brescia, Brescia
  - University ""Magna Graecia"" Of Catanzaro, Catanzaro
  - Amyloidosis Research & Treatment Center, Fondazione Irccs Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Senese - Policlinico Santa Maria Alle Scotte, Siena
  - University of Torino, S. Anna Hospital- City of Health and Science, Torino
- Latvia (5):
  - ARS, Riga
  - Latvian Maritime Medicine Centre, Riga
  - N. Lietuviete Private Practice, Riga
  - Private Practice, Riga
  - RiGa 1st Hospital, Riga
- Lithuania (2):
  - Jsc Kardiolita, Vilnius
  - Medical Center Maxmeda, Vilnius
- Radboud Universitair Medical Center, Nijmegen, Netherlands
- Gabinet Lekarski Specjalistyczny "Sonus" Lemieszczuk Boguslaw, Warsaw, Poland
- Portugal (3):
  - Centro hospitalar do Baixo vouga, EPE, Aveiro
  - Private Practice, Coimbra
  - Clinica Jardim das Amoreiras, Lisbon
- Romania (4):
  - Centrul Medical Euromed, Bucharest
  - Genesys Fertility Center, Bucharest
  - Spitalul Clinic Dr. Ioan Cantacuzino, Bucharest
  - Elena Doamna Obstetrics and Gynecology Clinical Hospital, Iași
- Spain (20):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitario de Cruces, Barakaldo
  - ASSIR OSONA (Atencio a la Salut Sexual i Reproductiva) - ICS (Institut Catala de la Salut), Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General Hospitalet CSI, Barcelona
  - Hospital Universitari Quiron Dexeus Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Clinic de Nefrologia i Urologia - ICNU, Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario de Guadalajara (HUG), Guadalajara
  - Hospital Clinico San Carlos, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Instituto Palacios, Salud y Medicina de la Mujer, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Quironsalud Toledo, Toledo
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (2):
  - Danderyds Sjukhus AB, Stockholm
  - Karolinska Institutet, Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (18):
  - Royal United Hospital, Bath - Royal United Hospital Bath NHS Trust, Bath
  - Royal Bolton Hospital, Bolton
  - University Hospital of North Durham, Durham
  - London North West Healthcare NHS Trust, Harrow
  - Hull Royal Infirmary - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Hinchingbrooke Health Care NHS Trust - Hinchingbrooke Hospital, Huntingdon
  - Leicester General Hospital, Leicester
  - North Middlesex University Hospital, London
  - Queen Charlotte's & Chelsea Hospital, London
  - Royal Manchester Children's Hospital - Manchester University NHS Foundation Trust, Manchester
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - Royal Victoria Infirmary - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Norfolk and Norwich University Hospital, Norwich
  - Rosemere Cancer Centre - Royal Preston Hospital, Preston
  - Sheffield Teaching Hospitals NHS Foundation Trust - Jessop Wing, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospital Of North Tees - North Tees And Hartlepool Nhs Foundation Trust, Stockton-on-Tees
  - Royal Stoke University Hospital - University Hospital of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No